CLINICAL TRIAL: NCT06550024
Title: SakuraBead Used as Resorbable Embolic for Genicular Artery Embolization
Acronym: SURE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CrannMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CI570
Record Dates: First submitted 2024-08-07; First posted 2024-08-12 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Osteo Arthritis Knee; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases; Arthritis; Osteoarthritis
Keywords: Genicular Artery Embolization; GAE; Knee Embolization; Knee OA; Knee Osteoarthritis
MeSH Terms: conditions — Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases; Arthritis; Osteoarthritis; Osteoarthritis, Knee | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Genicular Artery Embolization (GAE) (Experimental): Temporary Embolization of Genicular Arteries using Resorbable Microspheres
  Interventions: Device: SakuraBead Resorbable Microspheres
- Corticosteroid Injection (Active Comparator): Corticosteroid injection in the knee
  Interventions: Drug: Corticosteroid Injection

INTERVENTIONS:
Device: SakuraBead Resorbable Microspheres — Temporary Embolization of Genicular Arteries using SakuraBead Resorbable Microspheres
  Arms: Genicular Artery Embolization (GAE)
Drug: Corticosteroid Injection — Corticosteroid injection in the knee
  Arms: Corticosteroid Injection

SUMMARY:
An open label, prospective, two-arm, multicenter, randomized controlled trial comparing SakuraBead genicular artery embolization (GAE) with a control (corticosteroid injection).

DETAILED DESCRIPTION:
To compare safety and efficacy of SakuraBead with corticosteroid injection for the treatment of pain secondary to knee osteoarthritis. Treatment will be performed on a total of approximately 89 patients who will be followed up for a period of 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is able and willing to provide written informed consent, and
2. Clinical diagnosis of knee OA, and
3. Moderate to severe knee pain (WOMAC Pain ≥ 10), and
4. Pain refractory to at least 3 months of conservative therapies (anti-inflammatory drugs, or physical therapy, or intra-articular injections), and
5. Kellgren-Lawrence grade 1, 2 or 3 on radiograph of the knee, and
6. Age ≥ 40 years and < 80 years, and
7. Able to comply with all treatments and follow-up visits.

Exclusion Criteria:

1. Severe knee OA (Kellgren-Lawrence grade 4), or
2. Current infection of target joint, or
3. Life expectancy less than 36 months, or
4. Known advanced atherosclerosis as defined by history of lower extremity or pelvis arterial bypass graft, lower extremity or pelvis arterial stent placement or prior history of vascular claudication, or
5. Rheumatoid or known serologic diagnosis of autoimmune arthritis, or
6. Prior knee replacement surgery in the target knee, or
7. Pain score of >3 NRS on the non-target knee, or
8. An acute internal derangement of the target knee, or
9. History of uncorrectable coagulopathy, or
10. Prior iodinated contrast reaction resulting in anaphylaxis, or
11. Active pregnancy as demonstrated by urine or serum β-hCG, or lactating female, or planning pregnancy in the following 12 months, or
12. Has undergone an invasive treatment (including but not limited to: corticosteroid injection, hyaluronic acid injections, nerve ablation) in the target knee within the past 3 months, or
13. Contraindication to MRI, or
14. At the discretion of the Principal Investigator

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Estimated)
Dates: Start 2024-11-28 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint - Proportion of Responders | 6 Months
  Compare the proportion of responders* (defined as ≥50% reduction in WOMAC Pain** score and ≥2 point reduction in NRS***) between the Investigational procedure and Control at 6 months.
  * Non-responders will include subjects experiencing device-related SAEs. **Western Ontario and McMaster Universities Osteoarthritis Pain Index. Scale: 0-20, where a lower score represents a better outcome ***NRS: Numeric Rating Scale that measures pain from 0 (no pain) to 10 points (worst pain).
Primary Safety Endpoint - Freedom from treatment-related SAEs | 6 Months
  Freedom from treatment-related serious adverse events (SAE) through 6 months following the index procedure (proportions will be compared between Investigational procedure and Control).

SECONDARY OUTCOMES:
Proportion of Responders at 1 Month and 3 Month | 1 Month and 3 Months
  Compare the proportion of responders* (defined as ≥50% reduction in WOMAC Pain** score and ≥2 point reduction in NRS***) between the Investigational procedure and Control at 1 Month and 3 Months.
  * Non-responders will include subjects experiencing device-related SAEs. **Western Ontario and McMaster Universities Osteoarthritis Pain Index. Scale: 0-20, where a lower score represents a better outcome ***NRS: Numeric Rating Scale that measures pain from 0 (no pain) to 10 points (worst pain).
Change in mean WOMAC Pain | 1 Month, 3 Months and 6 Months
  Compare mean change from baseline in the Western Ontario and McMaster University Osteoarthritis Index Pain (WOMAC Pain, Scale: 0-20, where a lower score represents a better outcome) between the Investigational procedure and Control at 1 Month, 3 Months and 6 Months.
Change in Numeric Rating Scale (NRS) | 1 Month, 3 Months and 6 Months
  Compare mean decrease in pain (measured using the Numeric Rating Scale (NRS)) between the Investigational procedure and Control at 1 month, 3 months and 6 months. Scale: 0-10, where a lower score means a better outcome.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (6):
  - University of Alabama Medicine, Birmingham, Alabama
  - Harbor UCLA Medical Center, Torrance, California
  - Advanced Vascular Institute, Panama City, Florida
  - IR Centers, Raleigh, North Carolina
  - Orthopedic and Fracture Specialists (O&FS), Portland, Oregon
  - IR Centers, Leesburg, Virginia
- Bokhua Memorial Cardiovascular Center, Tbilisi, Georgia
- Royal Berkshire NHS Foundation Trust, Reading, United Kingdom
- Nano Medical Clinic, Tashkent, Uzbekistan, Uzbekistan

IPD SHARING:
Plan to Share IPD: No